CLINICAL TRIAL: NCT01323413
Title: Determinants of Penumbra in Acute Ischemic Stroke Patients
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, rambam62, MD, Rambam Health Care Campus
Other Study IDs: 0080-11CTIL
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Acute Ischemic Stroke
Keywords: stroke; penumbra; determinants; CT perfusion
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- stroke: acute ischemic stroke patients

SUMMARY:
The purpose of the study is to examine the influence of demographic, clinical and laboratory characteristics on the presence and size of penumbra in acute ischemic stroke patients and to determine those of them which related significantly and independently to the presence and size of Penumbra. The examined factors will include demographic variables such as age, gender, ethnic background, vascular risk factors and medical history, clinical parameters such as time from stroke onset until arrival to the hospital, results of neurological evaluation by NIHSS and imaging findings, laboratory tests such as body temperature, blood pressure, glucose level, renal functions etc. and imaging findings - the presence and the size of collateral blood vessels, the state of carotid arteries (by CTA). The possible correlation between all this parameters and the presence and the size of penumbra as detected by CTP will be further examined.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke patients hospitalized in Rambam Health Care Campus between 2008-2010, and which have underwent neurological evaluation including NIHSS scale, Brain CT, CT angio and Ct perfusion.

Exclusion Criteria:

* Intracranial hemorrhage of any other brain condition

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: neurological ward
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2011-04; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Haifa, Israel